CLINICAL TRIAL: NCT01661387
Title: A European, Multi-Centre, Multi-Country, Post-Authorisation, Observational Study (Registry) of Patients With Chronic Adrenal Insufficiency (AI)
Brief Title: A European Post-Authorisation Observational Study (Registry) of Patients With Chronic Adrenal Insufficiency (AI)
Status: Terminated | Type: Observational
Why Stopped: Takeda submitted 900 patient years Interim Analysis to PRAC and requested study to be closed since primary objective had been fulfilled. PRAC agreed and on 17Sep2020 approved closure of EU-AIR Registry. Takeda announced study closure on 31Oct2020.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: 0918-400
Record Dates: First submitted 2012-08-06; First posted 2012-08-09 (Estimated); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Chronic Adrenal Insufficiency
Keywords: Adrenal insufficiency; DuoCort; Congenital adrenal hyperplasia (CAH); Modified release; Hydrocortisone
MeSH Terms: conditions — Adrenal Insufficiency; Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Plenadren: Modified release hydrocortisone
- Other Glucocorticoid Replacement Therapy

SUMMARY:
As a post-approval requirement of the European Medicines Agency, this European patient post authorization safety study is an observational study being conducted to monitor the safety of long-term treatment with Plenadren and other glucocorticoid replacement therapies in routine clinical practice in patients with chronic adrenal insufficiency (primary or secondary).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic adrenal insufficiency
* Written informed consent/assent in compliance with applicable country-specific and local regulations

Exclusion Criteria:

* Participation in an interventional clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic adrenal insufficiency (primary or secondary) who are receiving Plenadren or other glucocorticoid replacement therapies at endocrinology centres in certain European countries as part of their routine clinical care. Approximately 20 sites are planned for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 3258 (Actual)
Dates: Start 2012-08-07 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of intercurrent illness | approximately 10 years
  Monitor the safety of long-term treatment with PLENADREN and other glucocorticoid replacement therapies in patients with chronic AI
Incidence of adrenal crisis | approximately 10 years
  Monitor the safety of long-term treatment with PLENADREN and other glucocorticoid replacement therapies in patients with chronic AI
Incidence of serious adverse events | approximately 10 years
  Monitor the safety of long-term treatment with PLENADREN and other glucocorticoid replacement therapies in patients with chronic AI

CONTACTS AND LOCATIONS:
Overall Officials: Shire Director, Study Director — Shire
Locations (24):
- Germany (9):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Endokrinologiepraxis am Stuttgarter Platz, Berlin
  - Friedrich Alexander Universitat Erlangen Nurnberg, Erlangen
  - Universitätsklinikum Frankfurt, Frankfurt
  - LMU Klinikum der Universität München, München
  - Medicover Neuroendokrinologie, München
  - Medicover Oldenburg MVZ, Oldenburg
  - Endokrinologiezentrum Ulm Praxis, Ulm
  - Universitätsklinikum Würzburg, Würzburg
- Italy (3):
  - Università degli Studi Federico II, Napoli
  - Policlinico Umberto I, Rome
  - Policlinico Universitario Agostino Gemelli, Rome
- Netherlands (3):
  - Universitair Medisch Centrum Groningen, Groningen
  - Erasmus MC, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenborg
  - Universitetssjukhuset i Linköping, Linköping
- United Kingdom (7):
  - Queen Elizabeth Hospital, Birmingham
  - St James University Hospital, Leeds
  - Barts and The London NHS Trust, London
  - Royal Free Hospital, London
  - Christie Hospital, Manchester
  - Royal Victoria Infirmary, Newcastle
  - Churchill Hospital, Oxford

REFERENCES:
- [Derived] Ekman B, Quinkler M, Zhang P, Isidori AM, Murray RD, Wahlberg J; EU-AIR investigators. Mineralocorticoid effects of fludrocortisone and hydrocortisone in primary adrenal insufficiency: EU-AIR patient data. J Endocrinol Invest. 2025 Oct;48(10):2381-2392. doi: 10.1007/s40618-025-02657-7. Epub 2025 Sep 6. PMID 40913682
- [Derived] Quinkler M, Murray RD, Zhang P, Marelli C, Petermann R, Isidori AM, Ekman B. Characterization of patients with adrenal insufficiency and frequent adrenal crises. Eur J Endocrinol. 2021 May 4;184(6):761-771. doi: 10.1530/EJE-20-1324. PMID 33769953
- [Derived] Quinkler M, Ekman B, Zhang P, Isidori AM, Murray RD; EU-AIR Investigators. Mortality data from the European Adrenal Insufficiency Registry-Patient characterization and associations. Clin Endocrinol (Oxf). 2018 Jul;89(1):30-35. doi: 10.1111/cen.13609. Epub 2018 Apr 22. PMID 29682773
- [Derived] Murray RD, Ekman B, Uddin S, Marelli C, Quinkler M, Zelissen PM; the EU-AIR Investigators. Management of glucocorticoid replacement in adrenal insufficiency shows notable heterogeneity - data from the EU-AIR. Clin Endocrinol (Oxf). 2017 Mar;86(3):340-346. doi: 10.1111/cen.13267. Epub 2016 Dec 5. PMID 27801983
- [Derived] Ekman B, Fitts D, Marelli C, Murray RD, Quinkler M, Zelissen PM. European Adrenal Insufficiency Registry (EU-AIR): a comparative observational study of glucocorticoid replacement therapy. BMC Endocr Disord. 2014 May 9;14:40. doi: 10.1186/1472-6823-14-40. PMID 24884782
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fc34db2bf003ab459c7??page=1&idFilter=0918-400